CLINICAL TRIAL: NCT01303744
Title: A Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Tolerability of Multiple Dose Regimens of CHF 5074 and to Explore the Effects in Patients With Mild Cognitive Impairment
Brief Title: Evaluation of Safety & Tolerability of Multiple Dose Regimens of CHF 5074
Acronym: CT04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CERESPIR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1014-PR-0053; 2010-024270-19 (EudraCT Number)
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CHF 5074 1x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF 5074 1x
- CHF 5074 2x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF 5074 2x
- CHF 5074 3x (Experimental): oral tablet, multidose
  Interventions: Drug: CHF 5074 3x
- Placebo (Placebo Comparator): placebo, oral tablet, multidose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF 5074 1x — oral tablet, 1x, once a day in the morning for 12 weeks
  Arms: CHF 5074 1x
Drug: CHF 5074 2x — oral tablet, 1x, once a day in the morning for 4 weeks, followed by oral tablet, 2x, once a day in the morning for 8 weeks
  Arms: CHF 5074 2x
Drug: CHF 5074 3x — oral tablet, 1x, once a day in the morning for 4 weeks, followed by oral tablet, 2x, once a day in the morning for 4 weeks, followed by oral tablet, 3x, once a day in the morning for 4 weeks
  Arms: CHF 5074 3x
Drug: Placebo — oral tablet, once a day in the morning for 12 weeks
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of ascending oral doses of CHF 5074 administered once per day for up to 12 weeks to patients with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of amnestic or non-amnestic Mild Cognitive Impairment.
* Mini-Mental State Examination score higher than 24 at screening.
* MRI scan of the brain at screening with fluid-attenuation inversion recovery (FLAIR) and T2*-weighted gradient-recalled-echo (GRE) sequences.

Exclusion Criteria:

* Diagnosis of Alzheimer's disease according to the (DSM-IV-TR) or NINCDS-ADRDA criteria.
* Any medical condition that could explain the patients cognitive deficits.
* CT or MRI brain imaging results obtained within 12 months prior to baseline showing evidence of infection, infarction, or focal lesions of clinical significance
* MRI scan at screening showing more than 4 cerebral microhemorrhages (lesions with diameter ≤ 10 mm).
* Geriatric Depression Scale (30-point scale) score > 9 at screening.
* History of stroke.
* Modified Hachinski ischemic scale score > 4 at screening.
* Women of childbearing potential.
* Vitamin B12 or folate deficiency.
* Diagnosis of schizophrenia or recurrent mood disorder (including unipolar and bipolar disorders) within 3 years of screening.
* Current diagnosis of peptic ulcer or gastrointestinal bleeding within the last year and/or chronic inflammatory bowel disease.
* Concomitant use of donepezil at doses > 5 mg/day or other cholinesterase inhibitors (rivastigmine or galantamine) at any dose.
* Concomitant use of memantine at dose > 20 mg/day.
* Concomitant use of psychoactive drugs (sedatives, hypnotics, etc).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel S. Ross, MD, Principal Investigator — Memory Enhancement Center of America, Inc.; Gabriella Bottini, Prof., Principal Investigator — Osp. Niguarda Ca Granda
Locations (9):
- United States (5):
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Memory Center of New Jersey, Inc., Monroe Twp, New Jersey
  - Memory Enhancement Center of NJ, Inc., Toms River, New Jersey
  - Senior Adults Specialty Research, Austin, Texas
- Italy (4):
  - Clinica Santa Maria, Div Neurologia, Castellanza
  - Osp. Maggiore Policlinico, Clin. Neurol, Milan
  - Osp. Niguarda Ca'Granda, Dip. Di Neuroscienze, Milan
  - Nuovo Osp Civ S. Agostino Estense, Dip di Neuroscienze, Modena

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHF 5074 1x | CHF 5074 2x | CHF 5074 3x | Placebo
Started | 24 | 24 | 24 | 24
Completed | 24 | 24 | 24 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHF 5074 1x | CHF 5074 2x | CHF 5074 3x | Placebo | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.1) | 68.9 (8.5) | 69.0 (9.2) | 68.1 (8.0) | 68.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 11 | 8 | 40
  Male | 14 | 13 | 13 | 16 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 23 | 22 | 24 | 23 | 92
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 19 | 24 | 91
  Italy | 0 | 0 | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Differences in ∆sCD40L Levels Between CHF 5074 Doses and Placebo at Any Specific Time Point
Description: To assess if there were differences in ΔsCD40L levels between CHF 5074 doses and placebo
Time Frame: up to 12 weeks
Population: ITT
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | CHF 5074 1x | CHF 5074 2x | CHF 5074 3x | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
pg/ml | 270.28 (371.09) | 403.22 (377.79) | -1293.42 (362.69) | 242.49 (361.32)

2. Secondary Outcome: Measurement of Trough CHF 5074 Plasma Levels
Description: evaluate the pharmacokinetics (PK) of CHF 5074 in patients with MCI.
Time Frame: Days 85
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CHF 5074 1x | CHF 5074 2x | CHF 5074 3x | Placebo
Number analyzed (Participants) | 24 | 20 | 20 | 0
ng/ml | 5497 (4940) | 7882 (8231) | 19999 (17474) |

3. Secondary Outcome: Changes in Plasma ΔTNFα Concentrations
Time Frame: 29 days
Population: ITT
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | CHF 5074 1x | CHF 5074 2x | CHF 5074 3x | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
pg/ml | 2.57 (1.1) | -0.339 (1.09) | -1.568 (1.05) | 0.039 (1.05)

ADVERSE EVENTS:
Time Frame: Trial duration
Arm/Group | CHF 5074 1x | CHF 5074 2x | CHF 5074 3x | Placebo
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/24 | 1/24 | 1/24
Other Adverse Events (participants affected / at risk) | 9/24 | 18/24 | 11/24 | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF 5074 1x (N=24) | CHF 5074 2x (N=24) | CHF 5074 3x (N=24) | Placebo (N=24)
intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Acute congestive heart failure (Cardiac disorders) | 0 | 0 | 1 (1) | 0
cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 | 0 | 0
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
cerebrovascular accident (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
femur fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
adenocarcinoma f transverse colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF 5074 1x (N=24) | CHF 5074 2x (N=24) | CHF 5074 3x (N=24) | Placebo (N=24)
diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (7) | 5 (5) | 2 (2)
back pain (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 3 (4) | 1 (1)
headache (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (4)
nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (5) | 0 (0) | 0 (0) | 1 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No